CLINICAL TRIAL: NCT04644302
Title: Circulatory and Endothelial Coherence in COVID-19 and Non-COVID-19 Patients With Sepsis - Prospective, Observational Pilot Study
Brief Title: Circulatory Coherence in COVID-19 and Non-COVID-19 Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Vladimir Cerny, professor, University Hospital Hradec Kralove
Other Study IDs: FNHK_IGS_8144
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Viral Pneumonia; Sepsis
Keywords: microcirculation; endothelial glycocalyx; COVID-19
MeSH Terms: conditions — Pneumonia, Viral; Sepsis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-COVID sepsis: Patients admitted to ICU with sepsis of non-COVID origin
  Interventions: Diagnostic Test: microcirculation recording
- COVID sepsis: Patients admitted to ICU with sepsis of COVID origin
  Interventions: Diagnostic Test: microcirculation recording

INTERVENTIONS:
Diagnostic Test: microcirculation recording — non-invasive recording of sublingual microcirculation and blood sampling together with regular withdraws
  Other Names: biochemical markeres investigation

SUMMARY:
This prospective observational pilot study investigates circulatory coherence in patients with COVID and non-COVID sepsis by comparison of microcirculation, endothelial glycocalyx, and clinical course

DETAILED DESCRIPTION:
This prospective observational pilot study investigates circulatory coherence in patients with COVID and non-COVID sepsis by comparison of microcirculation (sublingual area video recordings and biochemical parameters of endothelial cells activation and damage) endothelial glycocalyx (sublingual area video recordings and biochemical parameter of glycocalyx degradation), and clinical course.

ELIGIBILITY:
Inclusion Criteria:

* adult
* ICU admission due to sepsis with organ failure
* need for organ support therapy (mechanical ventilation, CRRT, ECMO)
* clinical and/or laboratory signs of circulatory instability

Exclusion Criteria:

* family withdrawal/disagreement
* death within three days from ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU with signs of circulatory instability with any method of organ support. Patients expected to have a particular method of organ support for at least 3 days.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
change in Proportion of Perfused Vessels (PPV) parameter | 1st, 2nd and 3rd day
  PPV describes microcirculation dysfunction
change in Syndecan-1 serum concentration | 1st, 2nd and 3rd day
  Syndecan-1 is a marker of endothelial glycocalyx

SECONDARY OUTCOMES:
change in albuminuria | 1st, 2nd and 3rd day
  albuminuria is a marker of glomerular endothelial cells dysfunction
mortality in 28 days | 30 days
  mortality in 28 days from ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Třebeš, Czechia